CLINICAL TRIAL: NCT06784752
Title: A Phase III Multi-center, Randomized, Open-label Study to Evaluate the Efficacy and Safety of [177Lu]Lu-DOTA-TATE in Patients Newly Diagnosed With Grade 1 and Grade 2 (Ki-67 <10%) Advanced GEP-NET With High Disease Burden (NETTER-3)
Brief Title: Study to Evaluate the Efficacy and Safety of [177Lu]Lu-DOTA-TATE in Patients With Grade 1 and Grade 2 Advanced GEP-NET
Acronym: NETTER-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA601A62301; 2024-518325-15-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2024-12-19; First posted 2025-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Somatostatin Receptor Positive (SSTR+); Gastroenteropancreatic Neuroendocrine Tumor (GEP-NET)
Keywords: SSTR+; GEP-NET; Ki-67 <10%; AAA601; [177Lu]Lu-DOTA-TATE; newly diagnosed; well differentiated; advanced GEP-NETs; high disease burden; NETTER-3; Grade 1; Grade 2; Tumor-targeted radioligand therapy; RLT; octreotide LAR; Gastroenteropancreatice Neuroendocrine Tumor; PFS; Quality of life (QOL)/PRO; QoL; neuroendocrine tumor(s); Lutathera; Lutetium dotatate; Lutetium oxodotreotide
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Lymphoma, Follicular | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [177Lu]Lu-DOTA-TATE + Octreotide LAR (Experimental): Participants in this arm will receive [177Lu]Lu-DOTA-TATE plus Octreotide long-acting release (LAR).
  Interventions: Radiation: [177Lu]Lu-DOTA-TATE; Drug: Octreotide LAR
- Octreotide LAR (Active Comparator): Participants in this arm will receive Octreotide LAR only.
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Radiation: [177Lu]Lu-DOTA-TATE — [177Lu]Lu-DOTA-TATE will be administered 4 times during treatment period with frequency of every 8 weeks (Q8W)
  Arms: [177Lu]Lu-DOTA-TATE + Octreotide LAR
Drug: Octreotide LAR — Octreotide LAR will be administered Q8W when co-administered with [177Lu]Lu-DOTA-TATE in the investigational arm followed by Q4W.
  In the control arm Octreotide LAR will be administered Q4W.
  Other Names: SOM230

SUMMARY:
The purpose of the current study is to evaluate the efficacy and safety of [177Lu]Lu-DOTA-TATE plus octreotide long-acting release (LAR) versus octreotide LAR alone in newly diagnosed patients with somatostatin receptor positive (SSTR+), well differentiated Grade1 and Grade 2 (G1 and G2) (Ki-67 <10%) advanced gastroenteropancreatic neuroendocrine tumors (GEP-NETs) with high disease burden

DETAILED DESCRIPTION:
The study consists of a screening phase, a treatment phase and a follow-up phase. This study compares treatment with [177Lu]Lu-DOTA-TATE plus octreotide LAR and octreotide LAR only.

ELIGIBILITY:
Inclusion Criteria:

* Presence of metastasized or locally advanced, unresectable (curative intent), histologically proven, well differentiated Grade 1 or Grade 2 (Ki-67 <10%) gastroenteropancreatic neuroendocrine tumor (GEP-NET) diagnosed within 6 months prior to screening.
* Participants with high disease burden in the Investigator's opinion. Following criteria should be used as the guiding principle for determining high disease burden:

  * Primary tumor or a metastatic lesion > 4 cm
  * More than one tumor or metastatic lesions measuring > 2 cm
  * Elevated alkaline phosphatase > 2.5 X upper limit of normal (ULN)
  * Presence of bone metastasis
  * Presence of peritoneal metastasis
  * Symptoms due to tumor volume such as pain, fatigue, weight loss, anorexia etc.
  * Symptoms due to hormone excess requiring active management
  * Additionally, participants who, in the Investigator's opinion, have high disease burden due to their disease characteristics not specified above could also be considered eligible.
* Participants ≥ 12 years of age.
* RLI somatostatin receptor (SSTR) uptake on all target lesions (defined by RECIST v1.1 criteria) at least as high as normal liver uptake assessed within 3 months prior to randomization. Any of the RLI modalities as available (some examples are listed below) can be used as per local practice:

  * [68Ga]Ga-DOTA-TOC PET/CT or PET/MRI
  * [68Ga]Ga-DOTA-TATE PET/CT or PET/MRI
  * [64Cu]Cu-DOTA-TATE PET/CT or PET/MRI
  * Somatostatin receptor scintigraphy (SRS) (planar and/or SPECT/CT) with [111In]In-pentetreotide
  * SRS (planar and/or SPECT/CT) with [99mTc]Tc-octreotide.
* Adequate bone marrow and organ function as defined by the following laboratory values prior to receiving the first study treatment:

  * White blood cell (WBC) count ≥ 2 x 109/L
  * Platelet count ≥ 75 x 109/L
  * Hemoglobin (Hb) ≥ 8 g/dL
  * Creatinine clearance > 40 mL/min calculated by the Cockcroft Gault method
  * Total bilirubin ≤ 3 x ULN
  * Potassium within normal limits. Potassium level of up to 6.0 millimoles per liter (mmol/L) is acceptable at study entry if associated with creatinine clearance within normal limits calculated using Cockcroft-Gault formula. Mild decrease (grade 1) below lower limit of normal (LLN) is acceptable at study entry if considered not clinically significant by Investigator.
* ECOG performance status 0-1.
* Presence of at least 1 measurable site of disease.

Exclusion Criteria:

* Prior administration of a therapeutic radiopharmaceutical for GEP-NET at any time prior to randomization in the study.
* Any previous therapy with interferons, mTOR-inhibitors, chemotherapy or other systemic therapies except somatostatin analogues (SSAs) of GEP-NET. If as per Investigator's opinion a participant is candidate for such therapies, such participant must not be enrolled.
* Participant who received more than 4 cycles of prior SSAs (e.g., octreotide long-acting release) are not eligible. In addition, any participant receiving treatment with short-acting octreotide, which cannot be interrupted for 24 h before the administration of [177Lu]Lu-DOTA-TATE, or any participant receiving treatment with SSAs, which cannot be interrupted for at least 4 weeks before the administration of [177Lu]Lu-DOTA-TATE.
* Documented RECIST v1.1 progression during previous SSA treatments for the current GEP-NET at any time prior to randomization.
* Any previous radioembolization, chemoembolization and radiofrequency ablation for GEP-NET.
* Any major surgery within 12 weeks prior to randomization in the study.
* Known brain metastases.
* Participant with known intolerance to CT scans with intravenous (i.v.) contrast due to allergic reaction or renal insufficiency. If such a participant can be imaged with MRI, then the participant would not be excluded.
* Hypersensitivity to any somatostatin analogues, to the Investigational Medicinal Products (IMPs) active substance or to any of the excipients.
* Active severe urinary incontinence, severe voiding dysfunction, or urinary obstruction requiring an indwelling/condom catheter that, in the judgment of the Investigator, could prevent adhering to radiation safety instructions.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2030-09-27 (Estimated); Study Completion 2034-01-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) centrally assessed by Blinded Independent Review Committee (BIRC) | After observing approximately 88 PFS events as per BIRC assessments, expected after approximately 33 months from study start
  PFS is defined as the time from randomization to the first occurrence of progression (centrally assessed by Blinded Independent Review Committee (BIRC) according to RECIST v1.1) or death due to any cause.

SECONDARY OUTCOMES:
Time to Deterioration (TDD) (Key Secondary) | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  Time to deterioration is defined as the time from randomization to the first occurrence of a deterioration compared to the baseline scores or death from any cause for each of the following domains (tested separately) of EORTC QLQ-GI.NET21 [gastrointestinal scale (GI scale)] and EORTC QLQ-C30 questionnaires (fatigue, diarrhea, and global health scale).
Progression Free Survival (PFS) | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  PFS is defined as the time from randomization to the first occurrence of progression (Investigator assessed according to RECIST v1.1) or death due to any cause.
Objective Response Rate (ORR) | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  ORR: Rate of participants with best overall response (BOR) of partial response (PR) or complete response (CR) as per RECIST v1.1 (both Investigator and centrally assessed by BIRC).
Disease Control Rate (DCR) | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  DCR: Rate of participants with BOR of PR, CR or stable disease (SD) as per RECIST v1.1 (both Investigator and centrally assessed by BIRC).
Duration of Response (DOR) | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  DOR: The time from initially meeting the criteria for response (CR or PR) until the time of progression according to RECIST v1.1 or death due to underlying disease only.
Overall Survival (OS) | Until 60 month from randomization
  OS: Time from the randomization date until the date of death due to any cause.
Time to Deterioration (TDD) | At the time of primary PFS analysis after observing approximately 88 PFS events per BIRC assessment
  TTD is the time from randomization to the first occurrence of a deterioration compared to the baseline scores or death from any cause for EORTC QLQ-G.I.NET21 and EORTC QLQ-C30 domains not included among key secondary endpoints.
Absolute change from baseline in EORTC QLQ-G.I.NET21 domain | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  Quality of Life assessed by EORTC QLQ-G.I.NET21 (excluding GI scale) (domains not included as key secondary objectives)
Absolute change from baseline in the EQ-5D-5L index at each time point | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  Quality of Life assessed by EQ-5D-5L
Absolute change from baseline in EORTC QLQ-C30 domain | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start.
  Quality of Life assessed by EORTC QLQ-C30 (domains not included as key secondary objectives)
Dosimetry | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  Absorbed radiation dose in selected organs, tumor lesions and total body
Pharmacokinetic (PK) parameter: Area Under Curve (AUC) from [177Lu]Lu-DOTA-TATE blood radioactivity data | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1).
  The AUC from time zero to infinity (mass x time x volume-1)
PK parameter: Clearance from [177Lu]Lu-DOTA-TATE blood radioactivity data | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  Clearance is the total body clearance of drug from the plasma or blood (volume x time-1).
PK parameter: Distribution volume (Vz) from [177Lu]Lu-DOTA-TATE blood radioactivity data | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  The apparent volume of distribution during terminal phase (associated with λz) (volume)
PK parameter: half-life (T1/2) from [177Lu]Lu-DOTA-TATE blood radioactivity data | After observing approximately 88 PFS events as per BIRC assessment, expected after approximately 33 months from study start
  The elimination half-life associated with the terminal slope (λz) of a semi logarithmic concentration-time curve (time). Use qualifier for other half-lives

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (17):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - LSU Medical Center, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Piedmont Healthcare, Winston-Salem, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - TxO Austin Midtown, Austin, Texas
  - Texas Oncology, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Center, Wytheville, Virginia
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- France (6):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Italy (6):
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Utrecht, Netherlands
- Poland (5):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com